CLINICAL TRIAL: NCT02949739
Title: Lifestyle Intervention to Prevent Type 2 Diabetes Amongst South Asians With Central Obesity and Prediabetes
Brief Title: Prevention of Type 2 Diabetes Amongst South Asians With Central Obesity and Prediabetes
Acronym: iHealth-T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16SM3246
Record Dates: First submitted 2016-04-27; First posted 2016-10-31 (Estimated); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive lifestyle modification (Active Comparator): The investigators will recruit 3,600 South Asian men and women aged 40-70 years with i. central obesity (waist≥100 cm) and/or ii. prediabetes (HbA1c 6.0-6.4%) to the study (Index cases). Recruitment will be from the Indian subcontinent (India, Pakistan, Sri Lanka) and Europe (UK). Index cases will receive either i. intensive lifestyle modification (N=1,800); or ii. usual care (N=1,800).
  Intensive lifestyle modification follows clinically accepted, evidence based strategies to achieve >7% reduction in weight through improved diet and increased physical activity, and is delivered as 9 face-face and 13 telephone contact sessions over 12 months.
  Index cases will be followed for three years to identify new-onset T2D.
  Interventions: Behavioral: Intensive lifestyle modification
- Usual Care (No Intervention): The investigators will recruit 3,600 South Asian men and women aged 40-70 years with i. central obesity (waist≥100 cm) and/or ii. prediabetes (HbA1c 6.0-6.4%) to the study.
  Recruitment will be from the Indian subcontinent (India, Pakistan, Sri Lanka) and Europe (UK). Index cases will receive either i. intensive lifestyle modification (N=1,800); or ii. usual care (N=1,800).
  Usual care group will comprise one diabetes prevention session and written material.

INTERVENTIONS:
Behavioral: Intensive lifestyle modification — The intervention is delivered as 9 face-face and 13 telephone contact sessions over 12 months. Index cases are the focus for the intervention, but lifestyle modification encourages the whole family to adopt healthy living.
  Arms: Intensive lifestyle modification

SUMMARY:
The investigators' general goal is to identify approaches to risk stratification and health promotion through lifestyle modification that are acceptable, effective and efficient for prevention of T2D in South Asian communities from diverse settings.

DETAILED DESCRIPTION:
The specific aims of the proposed iHealth-T2D study are:

1. Determine whether intensive lifestyle modification vs usual care reduces risk of T2D (primary endpoint) amongst South Asians with i. central obesity; ii. prediabetes and iii. overall (with central obesity and / or obesity).
2. Investigate secondary endpoints, including health gains in family members. Identify social, demographic and environmental factors influencing primary and secondary endpoints.
3. Carry out a health economic analysis of lifestyle modifications vs usual care for prevention of T2D on the Indian subcontinent and Europe. Quantify the cost-effectiveness of screening by waist circumference vs HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference≥100cm OR HbA1c≥6.0%
* South Asian, Male or Female, and age 40-70 years

Exclusion Criteria:

* Known type 1 or 2 diabetes
* Fasting glucose≥7.0 mmol/L or HbA1c ≥6.5%
* Normal or underweight (body mass index<22kg/m2)
* Pregnant or planning pregnancy
* Unstable residence or planning to leave the area
* Serious illness
* Lack of capacity to consent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5244 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
>7% reduction in weight | 4 year
  The investigators aim to achieve this outcome by motivating study participants to improve diet habits and increase physical activity

SECONDARY OUTCOMES:
Reduction of ≥5 cm waist circumference | 4 year
  The investigators aim to motivate the participants to adopt a healthier lifestyle in order to achieve at least 5cm waist circumference reduction

CONTACTS AND LOCATIONS:
Overall Officials: John Chambers, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once the research is completed the data and results will be made fully anonymous (ie all personal information removed), and available for use by other researchers. Any remaining blood samples will be destroyed.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 2020
Access Criteria: According to Study Protocol

REFERENCES:
- [Derived] Muilwijk M, Loh M, Mahmood S, Palaniswamy S, Siddiqui S, Silva W, Frost GS, Gage HM, Jarvelin MR, Rannan-Eliya RP, Ahmad S, Jha S, Kasturiratne A, Katulanda P, Khawaja KI, Kooner JS, Wickremasinghe AR, van Valkengoed IGM, Chambers JC. The iHealth-T2D study: a cluster randomised trial for the prevention of type 2 diabetes amongst South Asians with central obesity and prediabetes-a statistical analysis plan. Trials. 2022 Sep 6;23(1):755. doi: 10.1186/s13063-022-06667-1. PMID 36068618
- [Derived] Kasturiratne A, Khawaja KI, Ahmad S, Siddiqui S, Shahzad K, Athauda LK, Jayawardena R, Mahmood S, Muilwijk M, Batool T, Burney S, Glover M, Palaniswamy S, Bamunuarachchi V, Panda M, Madawanarachchi S, Rai B, Sattar I, Silva W, Waghdhare S, Jarvelin MR, Rannan-Eliya RP, Gage HM, van Valkengoed IGM, Valabhji J, Frost GS, Loh M, Wickremasinghe AR, Kooner JS, Katulanda P, Jha S, Chambers JC. The iHealth-T2D study, prevention of type 2 diabetes amongst South Asians with central obesity and prediabetes: study protocol for a randomised controlled trial. Trials. 2021 Dec 18;22(1):928. doi: 10.1186/s13063-021-05803-7. PMID 34922608
- [Derived] Muilwijk M, Loh M, Siddiqui S, Mahmood S, Palaniswamy S, Shahzad K, Athauda LK, Jayawardena R, Batool T, Burney S, Glover M, Bamunuarachchi V, Panda M, Madawanarachchi M, Rai B, Sattar I, Silva W, Waghdhare S, Jarvelin MR, Rannan-Eliya RP, Wijemunige N, Gage HM, Valabhji J, Frost GS, Wickremasinghe R, Kasturiratne A, Khawaja KI, Ahmad S, van Valkengoed IG, Katulanda P, Jha S, Kooner JS, Chambers JC. Effects of a lifestyle intervention programme after 1 year of follow-up among South Asians at high risk of type 2 diabetes: a cluster randomised controlled trial. BMJ Glob Health. 2021 Nov;6(11):e006479. doi: 10.1136/bmjgh-2021-006479. PMID 34725039